CLINICAL TRIAL: NCT04310735
Title: Examining Brain Responses Linked to Emotion in Individuals Who Smoke Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephen Wilson, Associate Professor, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00011266; R21DA045853 (NIH)
Record Dates: First submitted 2020-03-11; First posted 2020-03-17 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Smoking, Tobacco
MeSH Terms: conditions — Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Expect-Yes (Experimental): Participants assigned to this condition will undergo a verbal smoking expectancy manipulation such that they will perceive an opportunity to smoke during the experimental session.
  Interventions: Behavioral: Verbal smoking expectancy manipulation
- Experimental: Expect-No (Experimental): Participants assigned to this condition will undergo a verbal smoking expectancy manipulation such that they will not perceive an opportunity to smoke during the experimental session.
  Interventions: Behavioral: Verbal smoking expectancy manipulation

INTERVENTIONS:
Behavioral: Verbal smoking expectancy manipulation — Instructions regarding whether or not participants will have an opportunity to smoke during the experimental session.

SUMMARY:
The study will use functional magnetic resonance imaging and facial coding methods to study individuals who smoke cigarettes. Smoking expectancy (the extent to which one perceives an opportunity to smoke a cigarette) will be manipulated using instructions, and the investigators will examine the effects of this manipulation on two primary endpoints under conditions designed to induce an urge to smoke: (1) brain responses measured using fMRI and (2) subjective affective responses measured using facial coding. Secondary endpoints include self-report measures of the desire to smoke and current affect.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be between the ages of 21 and 55.
* Participants must be right handed.
* Participants must be fluent English speakers.
* Participants must report smoking at least 6 cigarettes per day continuously for at least the 12 preceding months.
* Participants must have a baseline expired air carbon monoxide (CO) exceeding a cutoff based upon prior research in order to verify smoking status.

Exclusion Criteria:

* Individuals will be excluded if they report that they are actively trying to quit smoking.
* Individuals will be excluded if they report that they have had significant cardiovascular disease (such as heart disease, heart attack, stroke, or angina) or respiratory disease (such as asthma, chronic bronchitis, or COPD) during the past year.
* Individuals will be excluded if they report that they have used any of the following illicit substances more than 10 times in the previous 30 days: marijuana, cocaine, opiates such as heroin, methadone, benzodiazepines (such as Valium, Xanax), barbiturates, amphetamines, methamphetamines, PCP, LSD or any other hallucinogen.
* Individuals will be excluded if they report that they are currently taking prescription medications that previously have been found to affect blood flow responses in the brain.
* Individuals will be excluded if they have any known risk from exposure to high-field strength magnetic fields (e.g., pace makers), any irremovable metallic foreign objects in their body (e.g., braces), or a questionable history of metallic fragments that are likely to create artifact on the MRI scans.
* Individuals will be excluded if they meet criteria for current dependence on a substance other than nicotine based upon a brief structured interview.
* Individuals will be excluded if they report that they are not willing to refrain from using alcohol and recreational drugs for 24 hours and nicotine for 12 hours before the experimental lab visit.
* Individuals will be excluded if they currently use nicotine products other than cigarettes (e.g., chewing tobacco, snuff, e-cigarettes, or smoking cessation products).
* Individuals will be excluded if they are claustrophobic or are prone to becoming very uncomfortable in confined spaces.
* Individuals will be excluded if they report that they exclusively or primarily smoke "roll-your-own" cigarettes.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2019-10-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
De-identified data and related materials (e.g., scripts) will be made publicly available on the Open Science Framework (OSF) to facilitate replication. Similarly, unthresholded fMRI statistical maps will be made publicly available on NeuroVault.

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Testing: Participants asked to complete behavioral testing only during experimental session for initial piloting, to allow progress toward the aims of the project while research was initially shut down and then subsequently restricted due to the COVID-19 pandemic, and to troubleshoot technical challenges.
Period: Overall Study
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing
Started | 14 | 13 | 35
Completed | 13 | 9 | 27
Not Completed | 1 | 4 | 8
Not completed — Withdrawal by Subject | 1 | 3 | 8
Not completed — Equipment malfunction | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing | Total
Number analyzed (Participants) | 14 | 13 | 35 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 13 | 35 | 62
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.8 (9.6) | 31.7 (9.4) | 28.5 (7.3) | 30.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 23 | 33
  Male | 8 | 9 | 12 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 2 | 5
  Not Hispanic or Latino | 12 | 12 | 33 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 3 | 5 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 4 | 4
  White | 9 | 6 | 24 | 39
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 35 | 62
Annual Household Income [Count of Participants; unit: Participants]
  Less than $10,000 | 2 | 1 | 2 | 5
  Less than $15,000 ($10,000 to less than $15,000) | 1 | 0 | 2 | 3
  Less than $20,000 ($15,000 to less than $20,000) | 1 | 0 | 1 | 2
  Less than $25,000 ($20,000 to less than $25,000) | 2 | 3 | 6 | 11
  Less than $35,000 ($25,000 to less than $35,000) | 4 | 3 | 10 | 17
  Less than $50,000 ($35,000 to less than $50,000) | 2 | 3 | 3 | 8
  Less than $75,000 ($50,000 to less than $75,000) | 0 | 2 | 1 | 3
  $75,000 or more | 2 | 1 | 9 | 12
  Not reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Brain Activation During Smoking-related and Neutral Cues
Description: Blood-oxygen-level dependent (BOLD) signal measured using functional magnetic resonance imaging (fMRI) was analyzed as participants were presented with smoking-related and neutral cues. Following preprocessing with fMRIPrep (version 20.2.7), the FMRI Expert Analysis Tool (FEAT) from FMRIB's Software Library (FSL; version 6.0.7.4) was used to characterize brain activation differences in response to smoking-related versus neutral cues. Contrast of parameter estimate (COPE) values were calculated for each participant, and these COPE values were then extracted for two a priori regions of interest (ROIs) to compare activation patterns between the groups. Larger COPE values indicate greater differences in brain activation between smoking-related and neutral cues,
Time Frame: Approximately Day 7 (Visit 2)
Population: Participants who completed the scan session and who provided usable brain imaging data were included in analyses. Participants in the Behavioral Testing Arm did not complete a scan session and were not assessed for brain activation during smoking-related and neutral cues.
Measure: Mean (Standard Error); unit: contrast of parameter estimate
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No
Number analyzed (Participants) | 9 | 11
contrast of parameter estimate
  Ventromedial prefrontal cortex ROI (10-mm sphere centered at MNI x = -1, y = 46, z = -7) | 5.8 (2.4) | -1.6 (3.8)
  Dorsal anterior cingulate cortex ROI (10-mm sphere centered at MNI x = -2, y = 10, z = 38) | 1.1 (3.4) | -4.2 (2.8)
Statistical Analysis 1: Comparison: Experimental: Expect-Yes vs Experimental: Expect-No; The null hypothesis was that there is no difference in the population means of the two groups; Test type: Other — Independent-samples t-tests were conducted to compare the mean contrast of parameter estimate (COPE) values, derived from the contrast of smoking-related versus neutral cue activation, between the Expect-Yes and Expect-No groups in the ventromedial prefrontal cortex region of interest; p = 0.13, t-test, 2 sided — Statistical significance was defined a priori as p<0.05
Statistical Analysis 2: Comparison: Experimental: Expect-Yes vs Experimental: Expect-No; The null hypothesis was that there is no difference in the population means of the two groups; Test type: Other — Independent-samples t-tests were conducted to compare the mean contrast of parameter estimate (COPE) values, derived from the contrast of smoking-related versus neutral cue activation, between the Expect-Yes and Expect-No groups in the dorsal anterior cingulate cortex region of interest; p = .25, t-test, 2 sided — Statistical significance was defined a priori as p<0.05

2. Primary Outcome: Coded Facial Expressions Linked to Affect During Smoking-related and Neutral Cues
Description: Subjective affective responses were measured by using FaceReader software (version 9.1.7) to code the valence (positive or negative) of facial movements associated with emotional expression during the presentation of smoking-related and neutral cues. Possible values for valence range from -1 to 1, with higher values indicating greater positive affect,
Time Frame: Approximately Day 7 (Visit 2)
Population: Participants who provided usable facial expression data were included in analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing
Number analyzed (Participants) | 9 | 11 | 9
units on a scale
  Valence during smoking-related cues | -.27 (.09) | -.24 (.09) | -.23 (.08)
  Valence during neutral cues | -.27 (.10) | -.25 (.09) | -.18 (.08)
Statistical Analysis 1: Comparison: Experimental: Expect-Yes vs Experimental: Expect-No; The null hypothesis was that there is no difference in the population means of the two groups; Test type: Other — Independent-samples t-tests were conducted to compare mean valence values during smoking-related cues between the Expect-Yes and Expect-No groups; p = .80, t-test, 2 sided; Statistical significance was defined a priori as p<0.05
Statistical Analysis 2: Comparison: Experimental: Expect-Yes vs Experimental: Expect-No; The null hypothesis was that there is no difference in the population means of the two groups; Test type: Other — Independent-samples t-tests were conducted to compare mean valence values during neutral cues between the Expect-Yes and Expect-No groups; p = .87, t-test, 2 sided — Statistical significance was defined a priori as p<0.05

3. Secondary Outcome: Self-reported Urge to Smoke During Smoking-related and Neutral Cues
Description: Participants rated their urge to smoke during the presentation of smoking-related and neutral cues on a scale ranging from 1 (not at all) to 9 (extremely), with higher scores indicating a stronger desire to smoke. For each type of cue (smoking-related and neutral), repeated ratings were obtained across multiple trials. To report a single value for each Arm/Group, the ratings were averaged across all trials for each cue type.
Time Frame: Approximately Day 7 (Visit 2)
Population: Participants who provided usable ratings data were included in analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing
Number analyzed (Participants) | 9 | 11 | 9
units on a scale
  Self-reported urge during smoking-related cues | 7.4 (0.2) | 7.1 (0.6) | 6.3 (0.7)
  Self-reported urge during neutral cues | 4.9 (0.6) | 5.0 (0.6) | 3.7 (0.9)

4. Secondary Outcome: Self-reported Affect During Smoking-related and Neutral Cues
Description: Participants rated their current affect during the presentation of smoking-related and neutral cues on a scale ranging from 1 (very negative) to 9 (very positive), with higher scores indicating greater positive affect. For each type of cue (smoking-related and neutral), repeated ratings were obtained across multiple trials. To report a single value for each Arm/Group, the ratings were averaged across all trials for each cue type.
Time Frame: Approximately Day 7 (Visit 2)
Population: Participants who provided usable ratings data were included in analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing
Number analyzed (Participants) | 9 | 11 | 9
units on a scale
  Self-reported affect during smoking-related cues | 6.1 (0.3) | 5.5 (0.3) | 5.1 (0.7)
  Self-reported affect during neutral cues | 5.9 (0.2) | 5.4 (0.3) | 5.9 (0.3)

5. Secondary Outcome: Nicotine Dependence
Description: Participants' level of nicotine dependence was assessed using the total score on the Fagerström Test for Nicotine Dependence to help characterize the sample. Possible scores on the Fagerström Test for Nicotine Dependence range from 0 to 10, with higher scores indicating greater nicotine dependence.
Time Frame: Day 1 (Visit 1)
Population: Only participants with usable data for the specified outcome were included in the analysis (i.e., those with missing data were excluded).
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing
Number analyzed (Participants) | 14 | 13 | 17
units on a scale | 3.8 (0.6) | 4.1 (0.6) | 4.4 (0.3)

6. Secondary Outcome: Brain Activation During Positive and Negative Emotion Cues
Description: Blood-oxygen-level dependent (BOLD) signal measured using functional magnetic resonance imaging (fMRI) was analyzed as participants were presented with cues designed to elicit positive and negative emotion. Following preprocessing with fMRIPrep (version 20.2.7), the FMRI Expert Analysis Tool (FEAT) from FMRIB's Software Library (FSL; version 6.0.7.4) was used to characterize brain activation in response to positive and negative emotion cues. Contrast of parameter estimate (COPE) values were calculated for each participant, and these COPE values were then extracted for two a priori regions of interest (ROIs) to compare activation patterns between the groups. Larger COPE values indicate greater differences in brain activation between positive and negative emotion cues.
Time Frame: Approximately Day 7 (Visit 2)
Population: Participants who completed the scan session and who provided usable brain imaging data were included in analyses (i.e., those with missing data or unusable data due to quality issue such as excessive head motion were excluded). Participants in the Behavioral Testing Arm did not complete a scan session and were not assessed for brain activation during positive and negative emotion cues.
Measure: Mean (Standard Error); unit: contrast of parameter estimate
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No
Number analyzed (Participants) | 9 | 12
contrast of parameter estimate
  Ventromedial prefrontal cortex ROI (10-mm sphere centered at MNI x = -1, y = 46, z = -7) | 2.4 (5.9) | 5.5 (2.8)
  Dorsal anterior cingulate cortex ROI (10-mm sphere centered at MNI x = -2, y = 10, z = 38) | -10.8 (4.5) | -2.2 (5.2)

7. Secondary Outcome: Coded Facial Expressions Linked to Affect During Positive and Negative Emotion Cues
Description: Subjective affective responses were measured by using FaceReader software (version 9.1.7) to code the valence (positive or negative) of facial movements associated with emotional expression during the presentation of cues designed to elicit positive and negative emotion. Possible values for valence range from -1 to 1, with higher values indicating greater positive affect,
Time Frame: Approximately Day 7 (Visit 2)
Population: Participants who provided usable facial expression data were included in analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing
Number analyzed (Participants) | 9 | 12 | 19
units on a scale
  Valence during positive emotion cues | -.19 (.10) | -.17 (.10) | .03 (.05)
  Valence during negative emotion cues | -.24 (.10) | -.25 (.09) | -.12 (.04)

8. Secondary Outcome: Self-reported Urge to Smoke During Positive and Negative Emotion Cues
Description: Participants rated their urge to smoke during the presentation of cues designed to elicit positive and negative emotions on a scale ranging from 1 (not at all) to 9 (extremely), with higher scores indicating a stronger desire to smoke. For each type of cue (positive and negative emotion), repeated ratings were obtained across multiple trials. To report a single value for each Arm/Group, the ratings were averaged across all trials for each cue type.
Time Frame: Approximately Day 7 (Visit 2)
Population: Participants who provided usable ratings data were included in analyses. Participants in the Behavioral Testing Arm were not presented with cues designed to elicit positive and negative emotion (they were only presented with smoking-related and neutral cues) and therefore did not provide data for this secondary outcome.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No
Number analyzed (Participants) | 9 | 12
units on a scale
  Self-reported urge during positive emotion cues | 3.0 (.3) | 4.0 (.6)
  Self-reported urge during negative emotion cues | 6.1 (.5) | 5.8 (.4)

9. Secondary Outcome: Self-reported Affect During Positive and Negative Emotion Cues
Description: Participants rated their current affect during the presentation of cues designed to elicit positive and negative emotion on a scale ranging from 1 (very negative) to 9 (very positive), with higher scores indicating greater positive affect. For each type of cue (positive and negative emotion), repeated ratings were obtained across multiple trials. To report a single value for each Arm/Group, the ratings were averaged across all trials for each cue type.
Time Frame: Approximately Day 7 (Visit 2)
Population: Participants who provided usable ratings data were included in analyses.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing
Number analyzed (Participants) | 9 | 12 | 19
units on a scale
  Self-reported affect during positive emotion cues | 7.6 (.2) | 6.7 (.3) | 6.4 (.3)
  Self-reported affect during negative emotion cues | 2.8 (.3) | 2.9 (.3) | 3.7 (.3)

ADVERSE EVENTS:
Time Frame: Adverse data were collected for the duration of each of the two study visits, which were held an average of approximately 12 days apart.
Arm/Group | Experimental: Expect-Yes | Experimental: Expect-No | Behavioral Testing
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/13 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/35
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-20): https://cdn.clinicaltrials.gov/large-docs/35/NCT04310735/Prot_SAP_000.pdf